CLINICAL TRIAL: NCT03651466
Title: A First-in-Human, Single Ascending Dose, Phase 1, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Subcutaneously Administered GX-G6 in Male Healthy Volunteers.
Brief Title: Safety and Tolerability of GX-G6 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GX-G6_HV1
Record Dates: First submitted 2018-07-05; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: GX-G6 + placebo (Experimental): Single administration of pre-determined dose (Level I) GX-G6 (6 subjects) and pre-determined dose (Level I) placebo (2 subjects)
  Interventions: Drug: Gx-G6; Drug: Placebo
- Cohort 2: GX-G6 + placebo (Experimental): Single administration of pre-determined dose (Level II) GX-G6 (6 subjects) and pre-determined dose (Level II) placebo (2 subjects)
  Interventions: Drug: Gx-G6; Drug: Placebo
- Cohort 3: GX-G6 + placebo (Experimental): Single administration of pre-determined dose (Level III) GX-G6 (6 subjects) and pre-determined dose (Level III) placebo (2 subjects)
  Interventions: Drug: Gx-G6; Drug: Placebo
- Cohort 4: GX-G6 + placebo (Experimental): Single administration of pre-determined dose (Level IV) GX-G6 (6 subjects) and pre-determined dose (Level IV) placebo (2 subjects)
  Interventions: Drug: Gx-G6; Drug: Placebo
- (Optional) Cohort 5: GX-G6 + placebo (Experimental): Single administration of pre-determined dose (Level V) GX-G6 (6 subjects) and pre-determined dose (Level V) placebo (2 subjects)
  Interventions: Drug: Gx-G6; Drug: Placebo
- (Optional) Cohort 6: GX-G6 + placebo (Experimental): Single administration of pre-determined dose (Level VI) GX-G6 (6 subjects) and pre-determined dose (Level VI) placebo (2 subjects)
  Interventions: Drug: Gx-G6; Drug: Placebo

INTERVENTIONS:
Drug: Gx-G6 — Each subject will receive a single dose of either GX-G6 or placebo in randomized fashion.
Drug: Placebo — Each subject will receive a single dose of either GX-G6 or placebo in randomized fashion.

SUMMARY:
This study is a single-center, double-blind, placebo-controlled, phase I study with healthy male subjects receiving ascending single s.c. doses of GX-G6

DETAILED DESCRIPTION:
A screening examination will be performed within 28 days prior to dosing. Eligible subjects will return to the study center in the morning of Day -1 and will remain in-patient until discharge about 98 hours after dosing (after oral glucose tolerance test in the morning of Day 5) if there are no safety issues. The s.c. injection will be administered in the morning of Day 1. Ambulatory visits will take place on Days 7, 9 and 12. A follow-up visit will take place on Day 15 and a final visit on Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. male subjects aged between 18-50 years (both inclusive)
2. healthy subjects as determined by medical history, physical examination including vital signs, ECG and clinical laboratory testing
3. subjects who are able and willing to give written informed consent
4. male subjects must be using 2 acceptable methods for contraception (one of these methods should be a barrier method e.g. spermicide and condom) from start of dosing and refrain from fathering a child in the 3 months following dosing.

Exclusion Criteria:

History of:

1. clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing), especially allergy to macrolide antibiotics;
2. any clinically significant pancreatic, hepatic, renal, gastrointestinal, cardiovascular, respiratory, hematological, central nervous system diseases or other significant diseases which might influence either the safety of the subject or the absorption, metabolism or excretion of the active agent under investigation;
3. diabetes mellitus and thyroid dysfunction or other endocrine disorders;
4. malignancy;
5. substance abuse or addiction (alcohol, drugs) in the past 3 years.

   Present Condition:
6. participation in a clinical investigation within the 30 days prior to the planned first drug administration or during this trial;
7. participation in this study at a previous dose level;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence, nature and severity of Adverse events | Throughout 4 weeks of study
  All safety data will be evaluated descriptively

SECONDARY OUTCOMES:
Pharmacodynamics(PD) variables | Pre-dose and 24, 48, 72, 96, 144, 192, 264 and 336 hours after dosing
  Oral glucose tolerance test in mol/L
Pharmacokinetics(PK) variables | Pre-dose and 24, 48, 72, 96, 144, 192, 264 and 336 hours after dosing
  GX-G6 concentration in blood

CONTACTS AND LOCATIONS:
Overall Officials: mi-sun byun, Ph. D, Study Director — Genexine, Inc.
Locations (1):
- NUVISAN, Neu-Ulm, Germany